CLINICAL TRIAL: NCT06086158
Title: Effect of Reverse Nordic Exercise on Vertical Jump in Youth Soccer Players: Randomized Controlled Trial
Brief Title: Effect of Reverse Nordic Exercise on Vertical Jump in Youth Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Javier Reina Abellan, Doctor en Docencia e Innovación Educativa, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TFM2022
Record Dates: First submitted 2023-10-01; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Strength
Keywords: Soccer; Eccentric Force; Quadriceps; Reverse Nordic Hamstring Exercise; Vertical Jump

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator
Masking Description: The trial was open or unblinded, the nature of the intervention prevented it from being blinded from the participants. The investigator in charge of collecting the data and carrying out the statistical study was the blind evaluator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nordic Reverse Protocol (Experimental): The intervention group performed the reverse Nordic exercise or quadriceps drop protocol for four weeks in their training sessions. Participants assigned to the intervention group warm up for approximately 15/20 minutes, consisting of five minutes of continuous running at low speed (approximately 10 km/h), followed by 3 minutes of stretching the lower extremities and three separate progressive sprints.
  between them with two minutes of rest to finish, then they will carry out the corresponding series and repetitions of the protocol and continue with their usual training.
  Interventions: Procedure: Nordic Reverse Protocol
- Usual Training Sessions (No Intervention): The control group did not have any intervention, the participants randomly assigned to this group continued with their usual training sessions.

INTERVENTIONS:
Procedure: Nordic Reverse Protocol — The participant begins on their knees, with the trunk upright and fully aligned. At this moment, the soccer player slowly leans back, maintaining the starting position by means of a controlled flexion of the knees. This fall is executed at the lowest speed possible to maximize muscle load in the eccentric phase and reach the point of maximum flexion.
  Arms: Nordic Reverse Protocol

SUMMARY:
BACKGROUNDː The reverse nordic hamstring exercise is developed for the eccentric work of the rectus femoris. After performing Nordic exercise protocol (its original), the relationship between increased eccentric hamstring strength, improvements in sprint capacity and reduced incidence of injuries can be confirmed. The review of evidence, led us propose the relationship and the possible benefits that could exist in the performance of four weeks of reverse nordic exercise protocol and the vertical jump, measured with countermovement jump test (CMJ) on a platform of jump.

METHODSː An open randomized controlled trial was conducted, with an intervention and control group, to which they were randomly assigned. The sample was made of 19 players from the San Antonio de Murcia Catholic University Team in the youth A category, aged between 16 and 18 years old. The experimental group (n=10) performed the reverse nordic hamstring exercise protocol for four weeks, in addition to the usual training that they shared with the control group (n=9). Data collection for the CMJ test was done before starting the protocol and immediately after finishing it for all participants. Statistical analysis was carried out with the SPSS program.

ELIGIBILITY:
Inclusion Criteria:

* Between 16 and 18 years old
* Soccer Players

Exclusion Criteria:

* Pathologies or Musculoskeletal Injuries in the last 6 months
* Surgical Interventions in the lower extremities in the last 6 months

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Flight Time | It was performed 3 days after completing the 4-week reverse Nordic exercise protocol.
  Chronojump Boscosystem® contact platform (Barcelona), to measure the vertical jump (CMJ and Abalakov) and the Chronojump Boscosystem® Software version 1.7.1
Jump Height | It was performed 3 days after completing the 4-week reverse Nordic exercise protocol.
  Chronojump Boscosystem® contact platform (Barcelona), to measure the vertical jump (CMJ and Abalakov) and the Chronojump Boscosystem® Software version 1.7.1

CONTACTS AND LOCATIONS:
Locations (1):
- Lara Sánchez Torres, Torre del Mar, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No